CLINICAL TRIAL: NCT04175886
Title: Effects of Tofacitinib on Body Composition, Bone Mineral Density and Bone Marrow Adiposity in Patients With Rheumatoid Arthritis: the TOFAT Project
Acronym: TOFAT
Status: Terminated | Type: Observational
Why Stopped: Design has to been modified due to the results from ORAL Surveillance
Sponsor: University Hospital, Lille (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018_38; 2019-001159-37 (EudraCT Number)
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-05

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; tofacitinib; body composition; bone marrow adiposity; bone marrow density
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with rheumatoid arthritis: Patients with rheumatoid arthritis with an indication for tofacitinib: 5mgx2 per day
  Interventions: Drug: Tofacitinib
- Healthy subjects: Healthy subjects matched to cases (1:1) on age (±5 years), sex, and menopausal status for women and body mass index (BMI, ±3 kg/m²)

INTERVENTIONS:
Drug: Tofacitinib — Patients will be treated with tofacitinib
  Groups: Patients with rheumatoid arthritis

SUMMARY:
Inflammatory rheumatic diseases (IRD), such as rheumatoid arthritis, are characterized by adverse changes in body composition. Lean mass and bone mineral density are usually reduced while adiposity (total fat mass, visceral adiposity…) is increased in comparison with healthy controls. Many factors may influence the body composition of those patients such as aging, Disease Modifying Anti-Rheumatic Drugs (DMARDs), nutrition and physical activity.

However, data on body composition and adverse changes under DMARDs in patients with rheumatoid arthritis (RA) are actually scarce. This is the case with tofacitinib (targeted synthetic DMARD or tsDMARD) while preliminary data let us think that this treatment may influence body composition and bone mineral density.

This study is going to be the first to focus on changes in body composition (fat mass and lean mass), bone mineral density and bone marrow adiposity under tofacitinib.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient's ≥18 years old with moderately to severely active Rheumatoid Arthritis (RA) (ACR/EULAR criteria )
* Previously untreated with Janus Kinase (JAK) inhibitors
* With an indication for tofacitinib will be eligible.
* All patients will have to be treated with tofacitinib either alone or with methotrexate. -Healthy volunteers should be ≥18 years old.

Exclusion Criteria:

* • treatment with more than three anti-Tumor Necrosis Factor alpha (TNFα). Patients who were receiving anti-TNFα will be required a washout period lasting at least five-half-lives before to start tofacitinib,

  * previously exposed to JAK inhibitors,
  * patients who were receiving non-anti-TNFα biologics (abatacept, tocilizumab, sarilumab or rituximab) will be required a washout period lasting at least five-half-lives before to start tofacitinib
  * Concomitant methotrexate (MTX) will be permitted if started ≥3 months prior to study start and at a stable dose (≤25 mg/week) for ≥4 weeks.
  * history or discovery of an osteoporotic fracture AND/OR T-score≤-3 if ≥50 years AND/OR Z-score ≤-3 if <50 years during the screening phase,
  * current treatment with oral corticosteroids higher than 10 mg prednisone/day,
  * pathologies or treatments that could affect the bone metabolism (breast cancer with aromatase inhibitors, gastrointestinal malabsorption, stomach cancer, primary hyperparathyroidism, uncontrolled hyperthyroidism…),
  * weight> 160 kg,
  * patients on restrictive diets or considering such a diet during the study period,
  * patients with an intense exercise program or planning to benefit from it during the study period,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is composed of adult patients with moderately to severely active RA for whom tofacitinib is indicated and who are followed in the department of rheumatology at Lille University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Variation in visceral adiposity (VAT or Visceral Adipose Tissue) in cm² | Between the measurement before and after 6 months of tofacitinib treatment (difference before/after).
  Variation in visceral adiposity (VAT or Visceral Adipose Tissue) in cm²

SECONDARY OUTCOMES:
Measurements of VAT in cm². | at baseline
  Measurements of VAT in cm²
Measurements of total fat mass (TBF) in kg, total lean mass (TLM) in kg, appendicular lean mass (aLM) in kg | at baseline
  Measurements of total fat mass (TBF) in kg, total lean mass (TLM) in kg, appendicular lean mass (aLM) in kg
Measurements of body fat percentage (%) | at baseline
  Measurements of body fat percentage (%)
Measurements of fat mass index (FMI) in kg/m² and skeletal muscle mass index (SMI) in kg/m² | at baseline
  Measurements of fat mass index (FMI) in kg/m² and skeletal muscle mass index (SMI) in kg/m²
Measurements of Bone mineral Density (BMD) in g/cm². | at baseline
  Measurements of Bone mineral Density (BMD) in g/cm².
Change in body fat percentage (% between measurement | Before and after 6 months of tofacitinib treatment (difference before/after).
  Change in body fat percentage (%) between measurement
Change in total fat mass (TBF) between measurement | Before and after 6 months of tofacitinib treatment (difference before/after).
  Change in total fat mass (TBF) in kg between measurement
Change in fat mass index (FMI) in kg/m², between measurement | Before and after 6 months of tofacitinib treatment (difference before/after).
  Change in fat mass index (FMI) in kg/m², between measurement
Change in total lean mass (TLM, kg) and appendicular lean mass (aLM) in kg between measurement | Before and after 6 months of tofacitinib treatment (difference before/after).
  Change in total lean mass (TLM, kg) and appendicular lean mass (aLM) in kg between measurement
Change in skeletal muscle mass index (SMI) in kg/m² between measurement | Before and after 6 months of tofacitinib treatment (difference before/after).
  Change in skeletal muscle mass index (SMI) in kg/m² between measurement
Change in BMD (in g/cm²) at the lumbar spine (L1-L4) and non-dominant total hip between measurement | Before and after 6 months of tofacitinib treatment (difference before/after).
  Change in BMD (in g/cm²) at the lumbar spine (L1-L4) and non-dominant total hip between measurement
Variation of bone remodelling markers (Cross-laps (CTX) and Type I procollagen N-terminal propeptide (P1NP)) between measurement | Before and after 6 months of tofacitinib treatment.
  Variation of bone remodelling markers (Cross-laps (CTX) and Type I procollagen N-terminal propeptide (P1NP)) between measurement
Variation in leptin (ng/ml) between measurement. | Before and after 6 months of tofacitinib treatment
  Variation in leptin (ng/ml) between measurement.
Change in bone marrow adiposity (%) at the lumbar spine between measurement | Before and after 6 months of tofacitinib treatment.
  Change in bone marrow adiposity (%) at the lumbar spine between measurement
Variation in Short Physical Performance Battery Protocol (SPPB) between measurement | Before and after 6 months of tofacitinib treatment.
  Variation in Short Physical Performance Battery Protocol (SPPB) between measurement
Changes in the parameters of the primary outcome and the secondary outcomes (n°2 to 8) | Before and after 12 months of tofacitinib treatment.
  Changes in the parameters of the primary outcome and the secondary outcomes (n°2 to 8)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Guillaume Letarouilly, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Lille University Hospital, Lille, France

REFERENCES:
- [Background] Dodington DW, Desai HR, Woo M. JAK/STAT - Emerging Players in Metabolism. Trends Endocrinol Metab. 2018 Jan;29(1):55-65. doi: 10.1016/j.tem.2017.11.001. Epub 2017 Nov 27. PMID 29191719
- [Background] Fleischmann RM, Huizinga TW, Kavanaugh AF, Wilkinson B, Kwok K, DeMasi R, van Vollenhoven RF. Efficacy of tofacitinib monotherapy in methotrexate-naive patients with early or established rheumatoid arthritis. RMD Open. 2016 Jul 26;2(2):e000262. doi: 10.1136/rmdopen-2016-000262. eCollection 2016. PMID 27493790
- [Background] Tatsumi Y, Nakao YM, Masuda I, Higashiyama A, Takegami M, Nishimura K, Watanabe M, Ohkubo T, Okamura T, Miyamoto Y. Risk for metabolic diseases in normal weight individuals with visceral fat accumulation: a cross-sectional study in Japan. BMJ Open. 2017 Jan 16;7(1):e013831. doi: 10.1136/bmjopen-2016-013831. PMID 28093438
- [Result] Book C, Karlsson MK, Akesson K, Jacobsson LT. Early rheumatoid arthritis and body composition. Rheumatology (Oxford). 2009 Sep;48(9):1128-32. doi: 10.1093/rheumatology/kep165. Epub 2009 Jul 13. PMID 19602478
- [Result] Haugeberg G, Uhlig T, Falch JA, Halse JI, Kvien TK. Bone mineral density and frequency of osteoporosis in female patients with rheumatoid arthritis: results from 394 patients in the Oslo County Rheumatoid Arthritis register. Arthritis Rheum. 2000 Mar;43(3):522-30. doi: 10.1002/1529-0131(200003)43:33.0.CO;2-Y. PMID 10728744
- [Result] Toussirot E, Mourot L, Dehecq B, Wendling D, Grandclement E, Dumoulin G; CBT-506. TNFalpha blockade for inflammatory rheumatic diseases is associated with a significant gain in android fat mass and has varying effects on adipokines: a 2-year prospective study. Eur J Nutr. 2014 Apr;53(3):951-61. doi: 10.1007/s00394-013-0599-2. Epub 2013 Oct 31. PMID 24173963
- [Result] Marouen S, Barnetche T, Combe B, Morel J, Daien CI. TNF inhibitors increase fat mass in inflammatory rheumatic disease: a systematic review with meta-analysis. Clin Exp Rheumatol. 2017 Mar-Apr;35(2):337-343. Epub 2016 Dec 13. PMID 27974099
- [Result] Engvall IL, Tengstrand B, Brismar K, Hafstrom I. Infliximab therapy increases body fat mass in early rheumatoid arthritis independently of changes in disease activity and levels of leptin and adiponectin: a randomised study over 21 months. Arthritis Res Ther. 2010;12(5):R197. doi: 10.1186/ar3169. Epub 2010 Oct 21. PMID 20964833
- [Result] Tournadre A, Pereira B, Dutheil F, Giraud C, Courteix D, Sapin V, Frayssac T, Mathieu S, Malochet-Guinamand S, Soubrier M. Changes in body composition and metabolic profile during interleukin 6 inhibition in rheumatoid arthritis. J Cachexia Sarcopenia Muscle. 2017 Aug;8(4):639-646. doi: 10.1002/jcsm.12189. Epub 2017 Mar 18. PMID 28316139
- [Derived] Letarouilly JG, Paccou J, Badr S, Chauveau C, Broux O, Clabaut A. Stimulatory Effect of Tofacitinib on Bone Marrow Adipocytes Differentiation. Front Endocrinol (Lausanne). 2022 Jul 6;13:881699. doi: 10.3389/fendo.2022.881699. eCollection 2022. PMID 35873000